CLINICAL TRIAL: NCT00710476
Title: Effect of the Number of Inseminated Spermatozoa on Subsequent Human Embryonic Development in Vitro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Prof. Dr. T D'Hooghe, University Hospital, Gasthuisberg, Leuven, Belgium
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dwille2
Record Dates: First submitted 2008-01-04; First posted 2008-07-04 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-01

CONDITIONS: Spermatozoa and Embryos
MeSH Terms: interventions — Insemination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Insemination of the oocytes with a lower concentration of spermatozoa.
  Interventions: Procedure: Insemination
- 2 (No Intervention): Insemination with a normal concentration of spermatozoa.

INTERVENTIONS:
Procedure: Insemination — Insemination with a lower concentration of spermatozoa: 150 000 spermatozoa/ml
  Arms: 1

SUMMARY:
In order to reach fertilization in the context of IVF, the presence of high concentrations of spermatozoa is associated with a higher degree of sperm metabolism and a higher concentration of sperm degradation products, which may adversely affect not only sperm and oocyte viability and the fertilization rate. The effect of a high concentration of sperm used for oocyte insemination appears also to be negative on embryo development (Dumoulin et al 1992*). If that is true, lowering the sperm concentration for oocyte insemination might improve embryo quality and result in a higher implantation rate per embryo. Therefore, we tested the hypothesis that the percentage of 8 cell-embryos on day 3 after IVF is significantly higher (40%) after insemination with a low sperm concentration (150 000/ml spermatozoa) than after insemination with a higher sperm concentration (30%; group 600 000/ml spermatozoa).

DETAILED DESCRIPTION:
1. BACKGROUND

   In human in-vitro fertilization procedures, oocytes are usually inseminated with concentrations that vary between 50 000 and 150 000 spermatozoa per ml fertilization medium. It has been shown that increasing the concentration of spermatozoa to >200 000 per ml, results in decreased fertilisation rates (66,7% in the group inseminated with 200 000 spermatozoa/ml versus 79,7% in the group inseminated with 10 000-90 000/ml; p<0,001) (Mahadevan and Trounson, 1984). These results were confirmed by another study (Diamond, Rogers et al., 1985). The reason for this decreased fertilisation rate is unclear but it has been speculated that the presence of high concentrations of sperm metabolism or degradation products associated with larger numbers of spermatozoa may adversely affect sperm and oocyte viability. Dumoulin et al. 1992 showed that increasing the sperm concentration affects not only the fertilisation rate but also the embryo development (Dumoulin, Bras et al., 1992). Significantly fewer fast-developing embryos (4-cell and 5- to 8-cell stages) were found on day 2 in the 100 000/ml group (53.4%) than in the 50 000/ml group (65.5%; p<0.05).

   At the Leuven University Fertility Centre (LUFC) oocytes have been inseminated traditionally for more than 15 years now with a higher sperm concentration (600 000/ml spermatozoa) than the average concentrations published (50 000 to 200 000 motile sperm/ml) (Chen and Kattera, 2006; Dumoulin, Bras et al., 1992; Racowsky, Combelles et al., 2003) This higher concentration for the insemination may be the cause of the lower rate of 8-cell embryos on day 3 observed at the LUFC when compared to the literature. At the LUFC only 20% of the embryos reach the 8-cell stage on day 3. In the literature the proportion of 8 cell embryos on Day 3 has been reported to be between 30 and 37% (Chen and Kattera, 2006;Racowsky, Combelles et al., 2003;Racowsky, Orasanu et al., 2005).

   In this prospective randomised trial we will test the hypothesis that embryo development can be improved by reducing the sperm concentration at insemination. This will be the first randomised trial showing the effect of inseminating with 600 000 spermatozoa/ml on the embryo development on day 3.
2. MATERIALS AND METHODS

   * Patients All patients with at least four oocytes will be included in this study. Furthermore, for inclusion in the study, the semen sample at the day of pick-up needs to have a total motility count after processing of at least 10 x 106 /ml. All ICSI patients will be excluded from this study.
   * Randomisation For each patient, all oocytes will be randomly assigned to the low insemination concentration (150 000/ml) or the high concentration (600 000/ml). The randomization will be done at the time of oocyte retrieval according to the principle "one here - one there".
   * Results from pilot study Before starting this prospective randomised trial, we have conducted a pilot study to check whether the fertilisation rate was not influenced by the reduction of the insemination concentration. 268 oocytes of 21 patients were included in this pilot study. Only patients with a good prognosis (defined as a fertilization rate of at least 70 % in the previous cycle and good sperm parameters: at least 10 x 106 motile spermatozoa per ml after processing and minimal 60% motile spermatozoa) were selected. At first, the insemination concentration was halved. The fertilisation rate didn't change significantly when we inseminated with 300 000 spermatozoa per ml instead of with 600 000 per ml (75, 9% versus 68,7%; p<0,05). In the second part of the pilot study the concentration was lowered to 150 000/ml. There was no decrease in fertilisation rate with the reduced number of spermatozoa (76,6% in the 150 000 group versus 83,6% in the 600 000 group; p<0,05). On day 2 a 10 percent increase in the number of good quality embryos was noticed (53,1% 4-cell embryos in the 150 000 group versus 42,6% in the 600 000 group; p<0,05). But on day 3 no difference in the number of good quality embryos was observed in this small group (32,7% in the 150 000 group versus 36,1% in the 600 000 group; p<0,05). This pilot study showed that lowering the sperm concentration for insemination does not reduce the fertilization rate, and may have a beneficial effect on embryo development but more patients need to be studied to confirm this trend
   * Sperm preparation Sperm samples are prepared using a density gradient centrifugation technique. The samples are loaded on an Isolate gradient and centrifuged at 1450 rpm for 20 minutes. The resulting pellet is washed twice by centrifugation. Afterwards, the pellet is resuspended in 0,75 ml fertilization medium. After counting the sample is diluted to a final concentration of 10 x 106 motile spermatozoa per ml (this is the concentration used for the high insemination group). For the low insemination group the sperm sample will be diluted again to a concentration of 2.5 x 106 motile spermatozoa per ml.
   * Embryo culture and transfer During the oocyte aspiration the oocytes will be divided in two groups. The oocytes are placed in 750 µl fertilization medium with a maximum of 5 oocytes. After incubation at 37°C, oocytes are inseminated by adding 30 µl of the sperm sample with either the low or the high concentration. Fertilization is evaluated 18-20h after the insemination. Embryo quality is evaluated on day 2, 3 and 5 (cleavage stage, morphology and symmetry). Depending on the number of fertilized oocytes and on the number of previous cycles, embryo transfer is performed on day 2, 3 or day 5. According to the transfer policy of the Belgian law (Koninklijk Besluit, 1 juli 2003), the best embryo(s) (based on cleavage stage, morphology and symmetry) are transferred into the uterus. On the day of transfer all surplus embryos of sufficient quality are cryopreserved.
   * Outcome variables and Power calculation The primary outcome variable of this study is the embryo development evaluated by the number of good quality embryos on day 2 and day 3 (in 7 or 8 cell stage). To test the hypothesis that the percentage of 7 to 8 cell-embryos in the group with the low insemination concentration (150 000/ml spermatozoa) is significantly higher (40%) than the percentage of the group with the high insemination concentration (30%), power calculation revealed that 299 embryos are needed in each group on day 3 (beta= 0.8 and alpha <0.05). Other outcome variables of this study are the fertilization rate, the incidence of polyspermy, pregnancy rate and implantation rate per transferred embryo.

ELIGIBILITY:
Inclusion Criteria:

* All patients with at laest 4 oocytes
* A sperm sample with a total motility count after processing of at least 1000 000 spermatozoa per ml

Exclusion Criteria:

* All ICSI cycles

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2006-08

PRIMARY OUTCOMES:
embryo quality | 36 hours

SECONDARY OUTCOMES:
implantation rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'Hooghe, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven